CLINICAL TRIAL: NCT06629103
Title: A Randomized, Double-blind Placebo-controlled Study in Healthy Subjects to Compare the Bioavailability of EPA + DHA From Two Microalgal Sources to One Fish Source
Brief Title: A Study in Healthy Subjects to Compare the Bioavailability of EPA + DHA
Acronym: GOBO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-5-12-GOBO
Record Dates: First submitted 2024-09-16; First posted 2024-10-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Optimal Absorption of Omega-3; Healthy
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- life's Omega 1035DS (Active Comparator)
  Interventions: Dietary Supplement: life's Omega 1035DS
- life'sTM Omega O3020DS (Active Comparator)
  Interventions: Dietary Supplement: life's Omega O3020DS
- MEG-3TM 1812 TG (Active Comparator)
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: life's Omega 1035DS — A natural triglyceride derived from microalgae with minimum 365 mg DHA, minimum 100 mg EPA, and minimum 520 mg/g DHA + EPA. Participants receive 600mg/d of omega-3 fatty acids from the microalgal oil.
  Arms: life's Omega 1035DS
Dietary Supplement: Fish Oil — Commercially available fish oil product MEG-3 1812 TG with a minimum 100 mg DHA/capsule, minimum 160 mg EPA/capsule, and minimum 300 mg/g DHA+EPA. Participants receive 600mg/d of omega-3 fatty acids from the fish oil.
  Arms: MEG-3TM 1812 TG
Other: Placebo — The placebo capsules will be a mixture of corn and soybean oils. Participants receive 600mg/d of omega-3 fatty acids from the corn/soy placebo.
  Arms: Placebo
Dietary Supplement: life's Omega O3020DS — A natural triglyceride derived from microalgae with minimum 210 mg DHA, minimum 300 mg EPA, and minimum 510 mg/g DHA + EPA. Participants receive 600mg/d of omega-3 fatty acids from the microalgal oil.
  Arms: life'sTM Omega O3020DS

SUMMARY:
This is a randomised, double-blind, parallel, placebo-controlled study in healthy subjects to compare the absorption of two microalgal formulations, to a fish oil and a placebo.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained before any trial related assessments are performed.
2. 2. Healthy adult females ages 18-64 who are neither pregnant nor breastfeeding or healthy adult males ages 18-64 at the time of consent.

   a. Female participants of child-bearing potential (females who are post-menopausal, i.e., when there has been no menstruation for a minimum of 12 months prior to screening, are considered not to be of child-bearing potential), who are not surgically sterilized, must have a negative pregnancy test at screening and be willing to practice one of the following appropriate contraceptive methods until the last visit: i. Sexual abstinence. ii. Oral contraceptives. iii. Trans dermal patches or depot injection of a progestogen drug (starting at least 4 weeks prior to product administration).

   iv. Intrauterine device (IUD), intrauterine system (IUS), subdermal implant, or vaginal ring (placed at least 4 weeks prior to product administration).

   Contraceptives must be effective before the randomization visit.
3. Participant's body mass index (BMI) must be between 18 and 30 kg/m2 (inclusive) and participant must weigh a minimum of 50 kg (110 lbs)
4. Intakes of EPA+DHA of less than 200mg per day based on the FFQ
5. Omega-3 Index less than 4%
6. Agree not to change current diet and exercise frequency or intensity during entire study period

Exclusion criteria:

1. Participant has any health conditions that would prevent from fulfilling the study requirements, put the participant at risk or would confound the interpretation of the study results as judged by the Investigator on medical history and routine laboratory test results.
2. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the participant or the validity of the study results.
3. More specifically, history or presence of diabetes, high triglycerides (>150 mg/dL), or high cholesterol (>200 mg/dL).
4. Has a clinically significant abnormal finding on the medical assessment, medical history, vital signs or clinical laboratory results at screening.
5. History or presence of allergic or adverse response to omega-3-acid ethyl esters or triglycerides (EPA or DHA), or related drugs, or sensitivity or allergy to fish or shellfish.
6. History of coagulation disorder or current anticoagulation therapy.
7. Has been on a significantly abnormal* diet, as deemed by the investigator, during the 4 weeks preceding the first dose of study medication. *an abnormal diet will be considered if the participant has elected to change to a more or less restricted diet of any description (e.g., change to or from a vegetarian, vegan, gluten-free, lactose-free, etc.) or significantly increases or decreases their daily caloric intake.
8. Has participated in another clinical trial (randomised participants only) within 30 days prior to the first dose of study medication.
9. Has used prescription medication (excluding oral contraceptive and hormonal replacement therapy) within 4 weeks of screening or OTC medication within 7 days before the first dose that may affect omega-3 absorption or any study outcomes. This may include, but is not limited to: high-dose NSAIDs, bile acid sequestrants, statins, GLP-1 receptor agonists, anticoagulants and anti-inflammatory drugs. Occasional ibuprofen, paracetamol and low-dose aspirin use is permitted.
10. Regular use (more than once per week) of omega-3 supplements (e.g., fish/krill/algae/flaxseed oil) within 2 months; or has consumed any omega-3 supplements or omega-3-rich foods (e.g., fortified products, or fatty fish >2x/week) within 14 days before the first dose.
11. Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
12. History of substance abuse or treatment (including more than 14 alcoholic drinks per week) within the past 2 years based on the judgement of the investigator.
13. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
14. Has increase bleeding from existing pathological conditions or anticipates surgery prior to, throughout, or within 1 week after study participation.
15. Has any dental appointment scheduled throughout or within 1 week after study participation.
16. Has had a transient ischemic attack (TIA) or stroke or is at high risk for recurrent ischemic events.
17. Has had or currently has lesions with a propensity to bleed (such as ulcers).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To compare the bioavailability of 600 mg/day of Omega-3 fatty acids (EPA+DHA) from two microalgal sources to a fish source by comparing the change from baseline in the sum level of EPA and DHA in plasma phospholipids across all treatments. | 6 weeks
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 6 between MEG-3, O1035DS and O3020DS and placebo as determined by Gas Chromatography (GC).

SECONDARY OUTCOMES:
To compare the bioavailability by 600mg/day of Omega-3 fatty acids by comparing the change from baseline in the sum level of EPA and DHA in plasma phospholipids across all treatments at the end of a 2, 4, and 6 week supplementation study. | 2, 4 and 6 weeks
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 2, 4, and 6 between MEG-3, O1035DS, O3020DS and placebo as determined by Gas Chromatography (GC).
To compare the bioavailability of 600mg/day of Omega-3 fatty acids by comparing the change from baseline in Omega-3 Index across all treatments at the end of a 6 week supplementation study. | 6 weeks
  The change in the Omega-3 Index (percent of EPA + DHA in red blood cell membranes) from baseline to week 6 between MEG-3, O1035DS, O3020DS and placebo as determined by Gas Chromatography (GC).
To compare the bioavailability of 600mg/day Omega-3 fatty acids by comparing the change from baseline in the plasma phospholipid levels across all treatments at week 2 and week 4 of supplementation. | 2 and 4 weeks
  The change in plasma phospholipids EPA+DHA µg/ml levels from baseline to week 2 and baseline to week 4 between MEG-3, O1035DS, O3020DS and placebo as determined by Gas Chromatography (GC).
To compare the changes from baseline in lipoprotein levels following consumption of the microalgal oils, fish oil or placebo at the end of a 6-week supplementation study. | 6 weeks
  The change in total cholesterol, HDL- and LDL-cholesterol and triglyceride levels from baseline to week 6 between MEG-3, O1035DS, O3020DS and placebo as determined by a clinical analyser.

OTHER OUTCOMES:
Additional endpoint 1 | 2, 4 and 6 weeks
  Change from baseline in plasma phospholipid EPA at weeks 2, 4 and 6 in MEG-3, O3020DS, 1035DS and placebo adjusted for intake level.
Additional endpoint 2 | 2, 4 and 6 weeks
  Change from baseline in plasma phospholipid DHA at weeks 2, 4 and 6 in MEG-3, O3020DS, 1035DS and placebo adjusted for intake level.
Additional endpoint 3 - Cytokines | Baseline and 6 weeks
  Exploratory parameters (Cytokines) at baseline and week 6 will be analysed using ELISA.
Additional endpoint 3 - neurotransmitters | Baseline and 6 weeks
  Exploratory parameters (neurotransmitters) at baseline and week 6 will be analysed using ELISA.
Additional endpoint 3 - specialized pro-resolving mediators | Baseline and 6 weeks
  Exploratory parameters (specialized pro-resolving mediators) at baseline and week 6 will be analysed using ELISA.
Additional endpoint 3 - PhenoAge Accel Index | Baseline and 6 weeks
  Exploratory parameters (PhenoAge Accel Index) at baseline and week 6. This is a metric calculated from phenotypic and chronological age, albumin, creatinine, alkaline phosphatase, glycated haemoglobin, WBC count, lymphocyte percentage, haemoglobin, red cell distribution width, MCV and, glucose).
Additional endpoint 3 - Aging clock (iAge) | Baseline and 6 weeks
  Exploratory parameters (Aging Clock) at baseline and week 6. This is a metric calculated from CXCL9, CCL11, CCL3, leptin, IL-1beta, IL-5, IFN-alpha, IFN-gamma, IL-4.
Additional endpoint 3 - PhenoAge Clock | Baseline and 6 weeks
  Exploratory parameters (PhenoAge Clock) at baseline and week 6. An epigenetic clock comprised of DNA methylation (DNAm) algorithms that combine information from measurements across the genome to quantify variations in biological versus chronological aging.
Additional endpoint 3 - Brain Health Score | Baseline and 6 weeks
  Exploratory parameters (Brain Health Score) at baseline and week 6. Brain health score derived from plasma proteomic and metabolomic biomarkers .
Safety Endpoint 1 | 6 weeks
  Screening and final visit clinical chemistry (electrolytes and liver function tests) and haematology (full blood counts) profiles will be assessed by clinical analyser.
Safety Endpoint 2 | 6 weeks
  Vital signs: Blood pressure (BP) will be assessed at screening, baseline and final visit.
Safety Endpoint 2 | 6 weeks
  Vital signs: Heart rate (HR) will be assessed at screening and final visit.
Safety Endpoint 2 | 6 weeks
  Vital signs: Body temperature will be assessed at screening and final visit.
Safety Endpoint 3 | Baseline to 6 weeks
  Anthropometric: Weight (kg) will be assessed at screening, baseline and the final visit.
Safety Endpoint 3 | 6 weeks
  Anthropometric: Waist-hip-ratio (WHR) will be assessed at screening and the final visit.
Safety Endpoint 4 | 6 weeks
  Adverse event (AE) listing will be collected.
Safety Endpoint 5 | 6 weeks
  Serious Adverse Event (SAE) will be reported to HREC, United BioSource Corporation (UBC) in Geneva, and the sponsor.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Birkett, Study Director — DSM Nutritional Products, Inc.
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided